CLINICAL TRIAL: NCT00586027
Title: Prospective Observational Study in Patients Undergoing Cardiac Surgery: Part 2: Is There a Correlation of Natriuretic Propeptide Type B With an Intraoperative Low Cardiac Output?
Brief Title: Is There a Correlation of Natriuretic Propeptide Type B With an Intraoperative Low Cardiac Output?
Status: Completed | Type: Observational
Sponsor: Klinikum Ludwigshafen (Other)
Responsible Party: Dr Andreas Lehmann, Klinikum der Stadt Ludwigshafen, Department of Anaesthesiology and Intensive Care Medicine
Other Study IDs: CI/NT-proBNP-12-2007
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Cardiac Surgery; Low Cardiac Output; Natriuretic Peptide B
Keywords: cardiac surgery; low cardiac output; natriuretic peptide B; mortality; morbidity
MeSH Terms: conditions — Cardiac Output, Low

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NT-proBNP: 150 consecutive patients undergoing cardiac surgery with an intraoperative measured cardiac output <2L/min/m².

SUMMARY:
Low output syndrome is a common complication in patients undergoing cardiac surgery. Its incidence was reported to be 2 to 6%. Morbidity and mortality of low output syndrome is high and the costs for treating the disease are immense.Natriuretic propeptide Type B (NT-proBNP) is a biological marker for the diagnosis, prognosis and therapy of cardiac failure after cardiac surgery.

Cardiac index and NT-proBNP will be correlated with morbidity and mortality. A critical threshold value for intraoperative cardiac index and NT-proBNP will be calculated.

DETAILED DESCRIPTION:
Low output syndrome is a common complication in patients undergoing cardiac surgery. Its incidence was reported to be 2 to 6% [1]. In patients suffering from low output syndrome cardiac output is severely reduced due to myocardial failure. Among other reasons for myocardial failure, ischemia, insufficient myocardial protection during aortic cross-clamping, and severely reduced ventricular function prior surgery are the most common risk factors for low output syndrome. Low output syndrome is treated with positive inotropic drugs and mechanical assist devices [2]. Morbidity and mortality of low output syndrome is high and the costs for treating the disease are immense.

If cardiac output cannot be increased cardiac failure persist and vital organs are hypoperfused. Critical and prolonged hypoperfusion results in single and multi organ failure. Until today a definite threshold for a critically reduced cardiac output or cardiac index requiring immediate therapy is not completely known. Cardiogenic shock is diagnosed by clinical signs and it is not diagnosed by cardiac output or cardiac index. The critical value for a severely reduces cardiac index was reported to be in a range of 1.75 to 2.5L/min/m² [3-5].

Natriuretic propeptide Type B (NT-proBNP) is a biological marker for the diagnosis, prognosis and therapy of cardiac failure after cardiac surgery [6,7].

The primary objective of this prospective observational study in 150 patients undergoing cardiac surgery with an intraoperative measured cardiac output <2L/min/m² is to monitor NT-proBNP for 7 days. Cardiac index and NT-proBNP will be correlated with morbidity and mortality [8]. A critical threshold value for intraoperative cardiac index and NT-proBNP will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient undergoing cardiac surgery
* Written informed consent
* Cardiac index before cardiopulmonary bypass <2L/min/m²

Exclusion Criteria:

* Missing consent
* Serum creatinine >1.5mg/dL [>123µmol/L]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 patients undergoing cardiac surgery, being monitored with a Swan-Ganz catheter and an intraoperatively before cardiopulmonary bypass measured cardiac index <2L/min/m².
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The primary objective is to monitor NT-proBNP for 7 days in patients with an intraoperative low cardiac output. Cardiac index and NT-proBNP will be correlated with morbidity and mortality. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Lehmann, MD, Principal Investigator — Klinikum der Stadt Ludwigshafen, Departement of Anesthesiology and Intensive Care Medicine
Locations (1):
- Klinikum der Stadt Ludwigshafen, Department of Anesthesiology and Intensive Care Medicine, Ludwigshafen, Germany

REFERENCES:
- [Background] Hausmann H, Potapov EV, Koster A, Krabatsch T, Stein J, Yeter R, Kukucka M, Sodian R, Kuppe H, Hetzer R. Prognosis after the implantation of an intra-aortic balloon pump in cardiac surgery calculated with a new score. Circulation. 2002 Sep 24;106(12 Suppl 1):I203-6. PMID 12354734
- [Background] Lehmann A, Boldt J. New pharmacologic approaches for the perioperative treatment of ischemic cardiogenic shock. J Cardiothorac Vasc Anesth. 2005 Feb;19(1):97-108. doi: 10.1053/j.jvca.2004.11.020. No abstract available. PMID 15747280
- [Background] Bohrer H, Schmidt H, Motsch J, Gust R, Bach A, Martin E. Gastric intramucosal pH: a predictor of survival in cardiac surgery patients with low cardiac output? J Cardiothorac Vasc Anesth. 1997 Apr;11(2):184-6. doi: 10.1016/s1053-0770(97)90211-1. PMID 9105990
- [Background] Hochman JS, Sleeper LA, Webb JG, Sanborn TA, White HD, Talley JD, Buller CE, Jacobs AK, Slater JN, Col J, McKinlay SM, LeJemtel TH. Early revascularization in acute myocardial infarction complicated by cardiogenic shock. SHOCK Investigators. Should We Emergently Revascularize Occluded Coronaries for Cardiogenic Shock. N Engl J Med. 1999 Aug 26;341(9):625-34. doi: 10.1056/NEJM199908263410901. PMID 10460813
- [Background] Adams HA, Baumann G, Gansslen A, Janssens U, Knoefel W, Koch T, Marx G, Muller-Werdan U, Pape HC, Prange W, Roesner D, Standl T, Teske W, Werner G, Zander R; I.A.G.-Schock. [Definition of shock types]. Anasthesiol Intensivmed Notfallmed Schmerzther. 2001 Nov;36 Suppl 2:S140-3. doi: 10.1055/s-2001-18174. German. PMID 11753724
- [Background] Cerrahoglu M, Iskesen I, Tekin C, Onur E, Yildirim F, Sirin BH. N-terminal ProBNP levels can predict cardiac failure after cardiac surgery. Circ J. 2007 Jan;71(1):79-83. doi: 10.1253/circj.71.79. PMID 17186982
- [Background] Provenchere S, Berroeta C, Reynaud C, Baron G, Poirier I, Desmonts JM, Iung B, Dehoux M, Philip I, Benessiano J. Plasma brain natriuretic peptide and cardiac troponin I concentrations after adult cardiac surgery: association with postoperative cardiac dysfunction and 1-year mortality. Crit Care Med. 2006 Apr;34(4):995-1000. doi: 10.1097/01.CCM.0000206110.94385.C4. PMID 16484891
- [Background] Polonen P, Ruokonen E, Hippelainen M, Poyhonen M, Takala J. A prospective, randomized study of goal-oriented hemodynamic therapy in cardiac surgical patients. Anesth Analg. 2000 May;90(5):1052-9. doi: 10.1097/00000539-200005000-00010. PMID 10781452